CLINICAL TRIAL: NCT01527786
Title: A Pilot Study of Functional Outcome in Postpartum Depression in Women Treated With Desvenlafaxine
Brief Title: Functional Outcome in Postpartum Depression in Women Treated With Desvenlafaxine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BC Women's Hospital & Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Shaila Misri, Dr., BC Women's Hospital & Health Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRISTIQ IOP # 3151A1-44
Record Dates: First submitted 2010-10-14; First posted 2012-02-07 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Depression
Keywords: Major Depressive Disorder, Postpartum Onset
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNRI treatment (Experimental): Participants are undergoing pharmacotherapy treatment with Desvenlafaxine (SNRI).
  Interventions: Drug: Desvenlafaxine

INTERVENTIONS:
Drug: Desvenlafaxine — 50mg-100mg everyday for 12 weeks over 7 study visits

SUMMARY:
Postpartum depressed women suffer from functional impairment in their mood, thoughts, cognition and physical well being leading to poor motivation, bonding difficulties, decreased productivity, conflict and neglect. Moderate/ severe depression responds best to a combination of antidepressants and counseling. This study will estimate the proportion of women who return to functionality after treatment with Desvenlafaxine and examine the differential impact of change in depression and anxiety symptoms on functionality over twelve weeks. Depression and anxiety symptoms will be monitored through six mood questionnaires; functional recovery will be monitored through a simple self-report questionnaire at each visit.

DETAILED DESCRIPTION:
Women will be recruited through a tertiary level care program and advertisements in BC Children's & Women's Hospital as well as St.Paul's Hospital, Vancouver, B.C., Canada. If deemed eligible for the study (meeting a diagnosis of postpartum depression with or without comorbid anxiety disorder) and the potential participant agrees to participate, consent will be signed. The participant will return on a bi-weekly basis for study visits, where mood and anxiety will be monitored, in addition to blood pressure and weight. Starting dose of Desvenlafaxine is 50mg, and this can be titrated to 100mg/per day if needed. Questionnaires will assess depression symptoms, anxiety symptoms, quality of life, panic disorder, obsessive-compulsive disorder and generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

1. To be able to read and write English.
2. Written informed consent before initiation of any study related procedures.
3. Diagnosis of Major Depressive Disorder (MDD) with onset of depressive symptoms within 12 months of delivery.
4. Diagnosis of additional comorbid panic, generalized anxiety or obsessive compulsive disorder, if they occur in addition to MDD.
5. Patients will be required to have a score of (greater than or equal than) 25 on the Montgomery-Asberg Depression Rating Scale (MADRS) at enrolment (moderate to severe depression).
6. Patients need to be referred by their usual treating primary care physician.
7. Those referrals must meet the clinic criteria for accepting referrals so that all potential participants are eligible to receive treatment in the clinic as per usual clinical practice.
8. Patient does not wish to pursue CBT elsewhere.
9. The patient is using an appropriate method of contraception, which may include abstinence, in order to avoid pregnancy during the study.
10. The patient is not currently breastfeeding.

Exclusion Criteria:

1. The patient is currently breastfeeding or pregnant.
2. The patient has a significant risk of suicide according to investigator's opinion or presents a score ³5 on item 10 (suicidal thoughts) of the MADRS.
3. The patient meets DSM-IV-TR criteria for:

   * current Post-traumatic Stress Disorder,
   * past or current manic or hypomanic episode,
   * past or current psychotic symptoms or disorder,
   * current drug or alcohol abuse or dependence,
   * current eating disorder (anorexia or bulimia).
4. The patient uses the following disallowed recent or concomitant medication within the specified time periods:

   * any antidepressant or any drug used for augmentation of antidepressant action within the last 1 week and 3 weeks for fluoxetine (longer half life) prior to baseline. Subject's mood will be monitored.
   * any hypnotics within the last week prior to baseline
   * oral antipsychotics within 2 weeks or depot antipsychotics within 6 months prior to baseline.
   * serotonergic medicinal products (for example, triptans, tryptophan, tramadol) within the last week prior to baseline.
   * Psychoactive herbal remedies (for example, St. Johns Wort, kava kava, valerian, ginkgo biloba) within the last 2 weeks prior to baseline.
   * any other drug with potential psychotropic effects within the last 2 weeks prior to baseline.
   * any anticonvulsant drug within the last 2 weeks prior to baseline.
   * any investigational product within 3 months prior to baseline.
5. The patient is currently receiving formal cognitive or behavioural therapy, systematic psychotherapy elsewhere, or plans to initiate such therapy during the study outside of the clinic.
6. The current depressive symptoms of the patient are considered by the investigator to have been resistant to two well-conducted antidepressant treatments of at least 6 weeks duration.
7. The patient has a serious illness or serious sequelae thereof, including liver or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological (including epilepsy), infectious, neoplastic, or metabolic disturbance. (If there is a history of such disease but the condition has been stable for at least one year and is judged by the investigator not to render inclusion unsafe and not to interfere with the patient's participation in the study, the patient may be included).

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Sheehan Disability Scale (SDS) | Baseline
  The Sheehan Disability Scale (SDS), which measures global functional impairment, as well as the individual score on each subscale (work/school; social life; family life/home responsibilities). To provide estimates for further studies, the mean change in score will be estimated with 95% confidence limits as a measure of variability. In addition, the proportion of subjects showing a change of more than clinically important change of more than 5 points will be estimated.
Sheehan Disability Scale (SDS) | 12 weeks
  The Sheehan Disability Scale (SDS), which measures global functional impairment, as well as the individual score on each subscale (work/school; social life; family life/home responsibilities). To provide estimates for further studies, the mean change in score will be estimated with 95% confidence limits as a measure of variability. In addition, the proportion of subjects showing a change of more than clinically important change of more than 5 points will be estimated.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS), the Hamilton Rating Scale- Anxiety (HAM-A), the Yale-Brown Obsessive Compulsive Scale (YBOCS), the Panic Disorder Severity Scale (PDSS), and the Penn Sate Worry Questionnaire (PSWQ). | Baseline
  Secondary efficacy assessment will be comprised of several measures. The secondary endpoint will be change from baseline on the total scores of these measures after 6 and 12-weeks of treatment. Resulting scores from these scales will be used to provide estimates and will be tabulated.
Montgomery-Asberg Depression Rating Scale (MADRS), the Hamilton Rating Scale- Anxiety (HAM-A), the Yale-Brown Obsessive Compulsive Scale (YBOCS), the Panic Disorder Severity Scale (PDSS), and the Penn Sate Worry Questionnaire (PSWQ). | 6 weeks
  Secondary efficacy assessment will be comprised of several measures. The secondary endpoint will be change from baseline on the total scores of these measures after 6 and 12-weeks of treatment. Resulting scores from these scales will be used to provide estimates and will be tabulated.
Montgomery-Asberg Depression Rating Scale (MADRS), the Hamilton Rating Scale- Anxiety (HAM-A), the Yale-Brown Obsessive Compulsive Scale (YBOCS), the Panic Disorder Severity Scale (PDSS), and the Penn Sate Worry Questionnaire (PSWQ). | 12 weeks
  Secondary efficacy assessment will be comprised of several measures. The secondary endpoint will be change from baseline on the total scores of these measures after 6 and 12-weeks of treatment. Resulting scores from these scales will be used to provide estimates and will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Shaila Misri, MD, Principal Investigator — BC Women's Hospital/UBC
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada